CLINICAL TRIAL: NCT02970253
Title: Direct Anterior Approach (DAA) for Total Hip Arthroplasty (THA): Capsular Resection Versus Capsular Flap Retention
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ZOL (Other)
Responsible Party: Principal Investigator, Jens Vanbiervliet, Resident Orthopedic Surgery, ZOL
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16/076U
Record Dates: First submitted 2016-11-03; First posted 2016-11-21 (Estimated); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Coxarthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Capsular resection (Active Comparator): Capsular resection
  Interventions: Procedure: Capsular resection
- Capsular retention (Active Comparator): Capsular retention
  Interventions: Procedure: Capsular retention

INTERVENTIONS:
Procedure: Capsular resection — Capsular resection
  Arms: Capsular resection
Procedure: Capsular retention — Capsular retention
  Arms: Capsular retention

SUMMARY:
Direct Anterior Approach (DAA) for Total Hip Arthroplasty (THA): Capsular resection versus capsular flap retention.

Prospective study design comparing clinical data in randomized THA patients who either had capsular resection or capsular flap retention.

ELIGIBILITY:
Inclusion Criteria:

* primary THA

Exclusion Criteria:

* neurologic disease
* painful contralateral THA
* severe back or knee pain
* rheumatology

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-11-11 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Clinical data will be measured with scoring list HHS (Harris Hip Score). | One year
  Hypothesis: No clinical difference in DAA using capsular resection vs retention. Clinical outcomes will be measured with scoring list HHS (Harris Hip Score).
Clinical data will be measured with scoring list WOMAC (The Western Ontario and McMaster Universities Arthritis Index). | One year
  Hypothesis: No clinical difference in DAA using capsular resection vs retention. Clinical outcomes will be measured with scoring list WOMAC (The Western Ontario and McMaster Universities Arthritis Index).
Clinical data will be measured with scoring list UCLA (University of California Los Angles activity score). | One year
  Hypothesis: No clinical difference in DAA using capsular resection vs retention. Clinical outcomes will be measured with scoring list UCLA ((University of California Los Angles activity score).
Clinical data will be measured with scoring list HOOS (Hip dysfunction and Osteoarthritis Outcome Score). | One year
  Hypothesis: No clinical difference in DAA using capsular resection vs retention. Clinical outcomes will be measured with scoring lists HOOS (Hip dysfunction and Osteoarthritis Outcome Score).

CONTACTS AND LOCATIONS:
Locations (1):
- ZOL, Genk, Limburg, Belgium